CLINICAL TRIAL: NCT04200638
Title: Effect of Three Mechanical Systems on Removal of Endotoxins From Necrotic Teeth With Apical Periodontitis After Two-visit RCT
Brief Title: Effect of Three Mechanical Systems on Removal of Endotoxins From Necrotic Teeth
Acronym: RCT2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, Dr. Jorge Paredes Vieyra DDS, MsC, PhD, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO2020
Record Dates: First submitted 2019-12-08; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: The trial design of this study will be a prospective, parallel, Randomized clinical trial (RCT).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, investigator and assessor.The trial design of this study will be a prospective, parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ProTaper Next group (Experimental): Clean and shape the necrotic canals with ProTaper instruments. In case of pain or inflammation 800mg Ibuprofen 3 times a day
  Interventions: Diagnostic Test: ProTaper Next
- WaveOne Gold group (Experimental): Clean and shape the necrotic canals with Wave One Gold instruments. In case of pain or inflammation 800mg Ibuprofen 3 times a day
  Interventions: Diagnostic Test: ProTaper Next

INTERVENTIONS:
Diagnostic Test: ProTaper Next — The canal fluid sample before and after will evaluate after root canal instrumentation

SUMMARY:
The patients will be randomly assigned into two equal groups Group : OneShape Group: ProtaperNext

Endodontics procedure steps:

Patient will be anesthetized by using infiltration local anesthesia or nerve block according to the tooth location in mandibular or maxillary arch respectively.

All caries will be removed, then isolation using rubber dam, the crown and surrounding structures will be disinfected with 30% H2O2( hydrogen peroxide) for 30 seconds, followed by 2.5% NaOCl for the same period of time and then inactivated with 5% sodium thiosulphate.

2- For the access cavity preparation, a sterile/apyrogenic high-speed diamond bur will be used in conjunction with manual irrigation with sterile saline. Before entering the pulp chamber, the access cavity will be disinfected according to the protocol described above.

2- Root canal length will be determined, by preoperative radiograph then (S1) will be taken by introducing a sterile/apyrogenic paper point #15/ 20 (5paper points) into the full length of the canal and left there for 1 minute. Then, the sample will be placed in an apyrogenic glass and stored in -20°. Then canal length will be confirmed by apex locator.

3- Cleaning and shaping will be done using either One shape or Protaper next rotary instruments in crown down preparation technique with the use of in an endodontic motor according to the manufacturer instructions, the canals will be thoroughly irrigated using 3ml of 2.5% Sodium hypochlorite between every subsequent instrument.

Lab procedures to identify microorganisms

DETAILED DESCRIPTION:
The patients will be randomly assigned into two equal groups Group : OneShape Group: ProtaperNext

Endodontics procedure steps:

Patient will be anesthetized by using infiltration local anesthesia or nerve block according to the tooth location in mandibular or maxillary arch respectively.

All caries will be removed, then isolation using rubber dam, the crown and surrounding structures will be disinfected with 30% H2O2( hydrogen peroxide) for 30 seconds, followed by 2.5% NaOCl for the same period of time and then inactivated with 5% sodium thiosulphate.

2- For the access cavity preparation, a sterile/apyrogenic high-speed diamond bur will be used in conjunction with manual irrigation with sterile saline. Before entering the pulp chamber, the access cavity will be disinfected according to the protocol described above.

2- Root canal length will be determined, by preoperative radiograph then (S1) will be taken by introducing a sterile/apyrogenic paper point #15/ 20 (5paper points) into the full length of the canal and left there for 1 minute. Then, the sample will be placed in an apyrogenic glass and stored in -20°. Then canal length will be confirmed by apex locator.

3- Cleaning and shaping will be done using either One shape or Protaper next rotary instruments in crown down preparation technique with the use of in an endodontic motor according to the manufacturer instructions, the canals will be thoroughly irrigated using 3ml of 2.5% Sodium hypochlorite between every subsequent instrument.

4-After root canal preparation, NaOCl will be inactivated with 5 mL of sterile 5% sodium thiosulphate for 1 minute, which then will be removed with 5 mL of sterile/apyrogenic saline solution., which then will be removed with 5 mL of sterile/apyrogenic saline solution. second endotoxin sample (S2) will be taken from the root canals. (5 paper point size of the master cone).

5- After completion of instrumentation and irrigation, obturation will be done using size 30/ 0.4 taper gutta-percha cones and auxiliaries as needed using the modified single cone technique.

Determination of Endotoxin Concentration Human endotoxin (ET) ELISA Kit will be used to measure endotoxin concentrations in the root canals before and after chemomechanical procedures.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion limitations were:

  1. nonappearance of radiographic proof of apical inflammation.
  2. irreversible pulpitis recognized by the positive reaction to thermal tests, and
  3. persistent pre-operative pain due to the pulpal condition.
  4. Patients must be in physical and emotional wellbeing.
  5. Any drug used seven days' previous study.

Exclusion Criteria:

1. impossibility to obtain patient's consent,
2. patients younger than 18 years. Necrotic teeth and teeth with periapical injury, root resorption,
3. Patients rejecting to join the research, those with issues with single-visit RCT, those consuming a specific kind of medicine such as painkillers or NSAIDs, and participants with some unrestrained systemic ailment were excluded too.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 to 65 years
Enrollment: 30 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-12-06 (Estimated)

PRIMARY OUTCOMES:
Endotoxin test for both groups | Endotoxin from fluid in ProTaper Next group
  measure endotoxin concentrations in the root canals before and after chemomechanical procedures. 24 hrs after root canal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Paredes Vieyra, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No
Clean and shape with two kinds of Ni-Ti instruments

REFERENCES:
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729